CLINICAL TRIAL: NCT00023452
Title: TBTC Study 26: Effectiveness and Tolerability of Weekly Rifapentine/Isoniazid for 3 Months Versus Daily Isoniazid for 9 Months for the Treatment of Latent Tuberculosis Infection
Brief Title: Three Months of Weekly Rifapentine and Isoniazid for M. Tuberculosis Infection
Acronym: PREVENT TB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3041; CDC TBTC Study 26 (Other: CDC TBTC)
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Tuberculosis
Keywords: Latent TB infection
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daily Isoniazid (Active Comparator): Isoniazid (INH) daily for 9 months (240 to 270 total doses).
  Interventions: Drug: Isoniazid (INH) daily for 9 months
- Weekly Isoniazid / Rifapentine (Experimental): Isoniazid / Rifapentine (RPT/INH) weekly for 3 months (11 to 12 total doses) given by Directly Observed Therapy (DOT)
  Interventions: Drug: RPT + INH once weekly for 3 months given by DOT

INTERVENTIONS:
Drug: RPT + INH once weekly for 3 months given by DOT — Rifapentine (RPT) 900 mg once-weekly x 12 doses (3 months) for persons > 50.0 kg. For persons < 50.0 kg, the following doses will be given (Weight/Dose): 10.0-14.0 kg / 300 mg; 14.1-25.0 kg / 450 mg; 25.1-32.0 kg / 600 mg; 32.1-50.0 kg / 750 mg.
  PLUS
  Isoniazid (INH) 15 mg/kg (rounded up to nearest 50 or 100 mg; 900 mg max) once weekly x 12 doses if > 12 years old. INH 25 mg/kg (round up to nearest 50 or 100 mg; 900 mg max) if 2-11 years old.
  Therapy will be given by Directly Observed Therapy (DOT).
  Other Names: INH; isoniazid; I; Rifapentine; RPT; P; Priftin; 3HP; 3INH/RPT
  Arms: Weekly Isoniazid / Rifapentine
Drug: Isoniazid (INH) daily for 9 months — Isoniazid (INH) 5 mg/kg (rounded up to nearest 50 or 100 mg; 300 mg max) daily x 270 doses (9 months) For children age 2 - 11, INH 10-15 mg/kg (round up to nearest 50 or 100 mg; 300 mg max) will be given.
  Other Names: Isoniazid; INH; I; 9INH
  Arms: Daily Isoniazid

SUMMARY:
Open-label, multi-center, Phase III clinical trial to compare the effectiveness and tolerability of a three-month (12-dose) regimen of weekly rifapentine and isoniazid (3RPT/INH) to the effectiveness of a nine-month (270-dose)regimen of daily isoniazid (9INH) to prevent tuberculosis (TB) among high-risk tuberculin skin-test reactors, including children and HIV-infected persons, who require treatment of latent TB infection (LTBI).

DETAILED DESCRIPTION:
The PRIMARY objective of this open-label Phase III clinical trial is to compare the effectiveness of a three-month (12-dose) regimen of weekly rifapentine and isoniazid (3RPT/INH) to the effectiveness of a nine-month (270-dose) regimen of daily isoniazid (9INH) to prevent tuberculosis (TB) among high-risk tuberculin skin-test reactors, including children and HIV-infected persons, who require treatment of latent TB infection (LTBI). The 3RPT/INH regimen will be given under direct observation and the 9INH regimen will be self-administered.

SECONDARY Objectives:

* Compare the rates of drug discontinuation due to adverse drug reactions associated with 3RPT/INH and 9INH.
* Compare the rates of drug discontinuation for any reason associated with 3RPT/INH and 9INH.
* Compare the rates of any grade 3, 4, or 5 drug toxicity associated with 3RPT/INH and 9INH.
* Compare treatment completion rates of 3RPT/INH and 9INH. Compare the efficacy (i.e., among persons who complete study-phase therapy) of 3RPT/INH and 9INH.
* Compare the effectiveness and tolerability of 3RPT/INH and 9INH in HIV-infected persons.
* Compare the effectiveness and tolerability of 3RPT/INH and 9INH in children < 18 years old.
* Compare the rates of methadone withdrawal associated with 3RPT/INH and 9INH among persons concomitantly receiving methadone.
* Describe patterns of antibiotic resistance among M. tuberculosis isolates in patients who develop TB despite treatment of latent infection.

Amendment of the study protocol to allow extension of enrollment to children < 12 years old and HIV-infected persons:

For assessment of the primary outcome, development of TB, a sample size of approximately 4,000 persons per arm will be required. To assess tolerability (one of the secondary outcomes) in sub-groups, children less than 12 years old and HIV-infected persons, a sample size of 644 per strata will be required. A sample size of 8,053 patients for the primary outcome was reached on February 15, 2008 (with expected follow-up completion time in 2010), leaving approximately 454 additional young children and 200 HIV-infected persons to be enrolled to achieve the targets of 644 for each group. The additional data on tolerability in those sub-groups will available for analysis in 2013.

ELIGIBILITY:
INCLUSION criteria:

* Males or nonpregnant, non-nursing females > 2 years old.
* Tuberculin (PPD) skin test reactors at high risk for developing TB but without evidence of active TB. High-risk reactors are defined as:

  1. Household and other close contacts of persons with culture-confirmed TB who are TST-positive as part of a contact investigation conducted within two years of the date of enrollment. Close contact is defined as > 4 hours in a shared airspace during a one-week period. Among close contacts, a positive TST is defined as > 5 mm induration after 5 TU of PPD placed intradermally using the Mantoux technique.
  2. TST converters--converting from a documented negative to positive TST within a two-year period. This is defined as persons with a tuberculin skin test of > 10 mm within two years of a nonreactive test or persons with an increase of > 10 mm within a two-year period.
  3. HIV-seropositive, TST positive (> 5 mm induration) persons.
  4. Persons with > 2 cm2 of pulmonary parenchymal fibrosis on chest X-ray, no prior history of TB treatment, > 5 mm induration on TST, and 3 sputum cultures negative for M. tuberculosis on final report.
* HIV-seropositive close contacts of persons with culture-confirmed TB, regardless of TST status. In addition, HIV-seropositive close contacts of persons with culture-confirmed TB who have a documented history of completing an adequate course of treatment for active TB or latent TB infection, are also eligible.
* Willing to provide signed informed consent, or parental consent and participant assent.

EXCLUSION criteria:

* Current confirmed culture-positive or clinical TB
* Suspected TB (as defined by the site investigator)
* Tuberculosis resistant to isoniazid or rifampin in the source case
* A history of treatment for > 14 consecutive days with a rifamycin or > 30 consecutive days with INH during the previous 2 years.
* A documented history of a completing an adequate course of treatment for active TB or latent TB infection in a person who is HIV-seronegative.
* History of sensitivity/intolerance to isoniazid or rifamycins
* Serum aminotransferase aspartate (AST, SGOT) > 5x upper limit of normal among persons in whom AST is determined
* Pregnant or nursing females
* Persons currently receiving or planning to receive HIV-1 protease inhibitors or nonnucleoside reverse transcriptase inhibitors in the first 90 days after enrollment.
* Weight < 10.0 kg

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8053 (Actual)
Dates: Start 2001-06; Primary Completion 2010-10 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elsa M Villarino, MD, MPH, Study Director — Centers for Disease Control and Prevention; Timothy Sterling, MD, Study Chair — Vanderbilt University Medical Center
Locations (26):
- United States (21):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - UCSD Medical Center, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Washington, D.C. VAMC, Washington D.C., District of Columbia
  - Emory University, Department of Medicine, Atlanta, Georgia
  - Chicago VA Medical Center (Lakeside), Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New Jersey Medical School, Newark, New Jersey
  - Columbia University/Presbyterian Medical Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Michael Debakey Veterans Affairs Medical Center, Houston, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Brazil
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Montreal Chest Institute McGill University, Montreal, Quebec
- Agencia de Salut Publica, Barcelona, Spain

REFERENCES:
- [Result] Sterling TR, Villarino ME, Borisov AS, Shang N, Gordin F, Bliven-Sizemore E, Hackman J, Hamilton CD, Menzies D, Kerrigan A, Weis SE, Weiner M, Wing D, Conde MB, Bozeman L, Horsburgh CR Jr, Chaisson RE; TB Trials Consortium PREVENT TB Study Team. Three months of rifapentine and isoniazid for latent tuberculosis infection. N Engl J Med. 2011 Dec 8;365(23):2155-66. doi: 10.1056/NEJMoa1104875. PMID 22150035
- [Derived] Moro RN, Mehaffy C, De P, Phillips E, Borisov AS, Sterling TR, Dobos KM. Assessment for Antibodies to Rifapentine and Isoniazid in Persons Developing Flu-Like Reactions During Treatment of Latent Tuberculosis Infection. J Infect Dis. 2024 Nov 15;230(5):1271-1278. doi: 10.1093/infdis/jiae180. PMID 38640958
- [Derived] Hedges KNC, Borisov AS, Saukkonen JJ, Scott NA, Hecker EJ, Bozeman L, Dukes Hamilton C, Kerrigan A, Bessler P, Moreno-Martinez A, Arevalo B, Goldberg SV. Nonparticipation reasons in a randomized international trial of a new latent tuberculosis infection regimen. Clin Trials. 2020 Feb;17(1):39-51. doi: 10.1177/1740774519885380. Epub 2019 Nov 6. PMID 31690107
- [Derived] Moro RN, Scott NA, Vernon A, Tepper NK, Goldberg SV, Schwartzman K, Leung CC, Schluger NW, Belknap RW, Chaisson RE, Narita M, Machado ES, Lopez M, Sanchez J, Villarino ME, Sterling TR. Exposure to Latent Tuberculosis Treatment during Pregnancy. The PREVENT TB and the iAdhere Trials. Ann Am Thorac Soc. 2018 May;15(5):570-580. doi: 10.1513/AnnalsATS.201704-326OC. PMID 29393655
- [Derived] Moro RN, Sterling TR, Saukkonen J, Vernon A, Horsburgh CR, Chaisson RE, Hamilton CD, Villarino ME, Goldberg S. Factors associated with non-completion of follow-up: 33-month latent tuberculous infection treatment trial. Int J Tuberc Lung Dis. 2017 Mar 1;21(3):286-296. doi: 10.5588/ijtld.16.0469. Epub 2017 Jan 13. PMID 28087928
- [Derived] Sterling TR, Scott NA, Miro JM, Calvet G, La Rosa A, Infante R, Chen MP, Benator DA, Gordin F, Benson CA, Chaisson RE, Villarino ME; Tuberculosis Trials Consortium, the AIDS Clinical Trials Group for the PREVENT TB Trial (TBTC Study 26ACTG 5259) The investigators of the TB Trials Consortium and the AIDS Clinical Trials Group for the PREVENT TB Trial are listed in the Supplement, item 17. Three months of weekly rifapentine and isoniazid for treatment of Mycobacterium tuberculosis infection in HIV-coinfected persons. AIDS. 2016 Jun 19;30(10):1607-15. doi: 10.1097/QAD.0000000000001098. PMID 27243774
- [Derived] Moro RN, Borisov AS, Saukkonen J, Khan A, Sterling TR, Villarino ME, Scott NA, Shang N, Kerrigan A, Goldberg SV. Factors Associated With Noncompletion of Latent Tuberculosis Infection Treatment: Experience From the PREVENT TB Trial in the United States and Canada. Clin Infect Dis. 2016 Jun 1;62(11):1390-1400. doi: 10.1093/cid/ciw126. Epub 2016 Mar 6. PMID 26951571
- [Derived] Sterling TR, Moro RN, Borisov AS, Phillips E, Shepherd G, Adkinson NF, Weis S, Ho C, Villarino ME; Tuberculosis Trials Consortium. Flu-like and Other Systemic Drug Reactions Among Persons Receiving Weekly Rifapentine Plus Isoniazid or Daily Isoniazid for Treatment of Latent Tuberculosis Infection in the PREVENT Tuberculosis Study. Clin Infect Dis. 2015 Aug 15;61(4):527-35. doi: 10.1093/cid/civ323. Epub 2015 Apr 22. PMID 25904367
- [Derived] Villarino ME, Scott NA, Weis SE, Weiner M, Conde MB, Jones B, Nachman S, Oliveira R, Moro RN, Shang N, Goldberg SV, Sterling TR; International Maternal Pediatric and Adolescents AIDS Clinical Trials Group; Tuberculosis Trials Consortium. Treatment for preventing tuberculosis in children and adolescents: a randomized clinical trial of a 3-month, 12-dose regimen of a combination of rifapentine and isoniazid. JAMA Pediatr. 2015 Mar;169(3):247-55. doi: 10.1001/jamapediatrics.2014.3158. PMID 25580725
- See also: (Click here for more information about the Tuberculosis Trials Consortium(TBTC) — https://www.cdc.gov/tb/research/tbtc.html?CDC_AAref_Val=https://www.cdc.gov/tb/topic/research/tbtc/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol design allowed enrollment of participants identified as members of the same household or group setting (such as group homes, settings) in clusters. The same treatment regimen to which a first participant was randomized could be assigned to other cluster members. All other participants enrolled were randomized individually.
Groups:
- 9INH: Participants who were high-risk tuberculin skin test (TST) reactors (household and other close contacts of active tuberculosis [TB] cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on chest x-ray [CXR], human immunodeficiency virus [HIV] infected participants) self-administered oral isoniazid (INH) tablets (aged greater than or equal to [≥12] years of age received 5 milligrams per kilogram [mg/kg] and participants 2-11 years of age received 10-15 mg/kg) once daily for 9 months (240 to 270 total doses).
- 3RPT/INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV-infected participants) received oral INH tablets (≥12 years of age received 15 mg/kg and participants 2-11 years of age received 25 mg/kg) and oral rifapentine (RPT) tablets (between 300-900 mg based on weight) once per week for 3 months (11 to 12 total doses) administered by Directly Observed Therapy (DOT), defined as a healthcare worker observing ingestion of each dose of RPT and INH.
Period: Overall Study
Arm/Group | 9INH | 3RPT/INH
Started | 3908 | 4145
Randomized | 3190 | 3174
Enrolled as Part of a Cluster | 718 | 971
Completed Treatment | 2585 | 3273
Not Treated | 149 | 105
Completed Study | 3174 | 3475
Completed | 2585 | 3273
Not Completed | 1323 | 872
Not completed — Ineligible for Study | 163 | 159
Not completed — Out of Window | 129 | 69
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 66 | 54
Not completed — Adverse Event | 139 | 196
Not completed — Lost to Follow-up | 293 | 60
Not completed — Physician Decision | 49 | 21
Not completed — Refused Treatment (continued follow-up) | 225 | 224
Not completed — Pregnant | 53 | 20
Not completed — Other | 204 | 69

BASELINE CHARACTERISTICS:
Groups:
- 9INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV infected participants) self-administered oral INH tablets (≥12 years of age received 5 mg/kg and participants 2-11 years of age received 10-15 mg/kg) once daily for 9 months (240 to 270 total doses).
- 3RPT/INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV infected participants) received oral INH tablets (≥12 years of age received 15 mg/kg and participants 2-11 years of age received 25 mg/kg) and oral RPT tablets (between 300-900 mg based on weight) once per week for 3 months (11 to 12 total doses) administered by DOT, defined as a healthcare worker observing ingestion of each dose of RPT and INH.
- Total: Total of all reporting groups
Arm/Group | 9INH | 3RPT/INH | Total
Number analyzed (Participants) | 3908 | 4145 | 8053
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [25 to 46] | 36 [25 to 47] | 35 [25 to 47]
Sex/Gender, Customized [Number; unit: participants]
  Female | 1812 | 1847 | 3659
  Male | 2096 | 2297 | 4393
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Rate of Culture-Confirmed TB Disease in Participants ≥18 Years of Age AND Culture-Confirmed or Probable (Clinical) TB Disease in Participants Less Than [<]18 Years of Age at 33 Months After Enrollment
Description: Cumulative TB disease rate defined as number of participants ≥18 years old with culture-confirmed TB disease (defined as positive culture for Mycobacterium tuberculosis [MTB]) and those <18 years old with probable (clinical) TB disease (defined as objective evidence of clinical TB disease [cough, fever, night sweats, weight loss, or hemoptysis] based on history or physical exam plus radiograph, computed tomography [CT] scan, other diagnostic tests PLUS response to antituberculosis therapy AND objective improvement of radiograph or other diagnostic tests; OR evidence of granuloma with organism positive for acid-fast bacilli [AFB], or caseating granulomata at autopsy or biopsy) between enrollment and the 990th Day of the Trial (33 months after enrollment, or end of the trial) per 100 participants with (w/)33 months of follow-up calculated using survival analysis methods (Kaplan-Meier approach).
Time Frame: Baseline up to Month 33
Population: Modified Intention-to-Treat (MITT) Population: all participants who enrolled in study and were eligible (Ineligible=source TB case resistant to INH or rifampin; source TB case culture-negative for MTB; positive TST not confirmed; MTB drug susceptibility test results not available for source TB case; or TB disease at enrollment).
Measure: Number; unit: TB cases per 100 participants w/followup
Groups:
- 9INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV infected participants) self-administered oral INH tablets (aged ≥12 years of age received 5 mg/kg and participants 2-11 years of age received 10-15 mg/kg) daily for 9 months (240 to 270 total doses).
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 3745 | 3986
TB cases per 100 participants w/followup | 0.43 | 0.19
Statistical Analysis 1: Comparison: 9INH vs 3RPT/INH; Test type: Non-Inferiority or Equivalence — The noninferiority test statistic was based on the difference of the nonparametric Kaplan-Meier estimators. The asymptotic variance of the test statistic was obtained through Greenwood's formula and a two-sided 95% confidence interval (CI) was constructed for the difference. If the upper bound of the CI was smaller than the noninferiority margin 0.75%, then the null hypothesis would be rejected and noninferiority could be claimed; Difference in Cumulative TB Disease Rate = -0.24, 95% CI 1-sided [upper limit 0.01] — The difference in cumulative TB disease rate is the rate in the 3RPT/INH arm minus the rate in the 9INH arm

2. Secondary Outcome: Cumulative Rate of Culture-Confirmed TB Disease in Participants ≥18 Years of Age AND Culture-Confirmed or Probable (Clinical) TB Disease in Participants <18 Years of Age at 24 Months Following Completion of Study Therapy
Description: Cumulative TB disease rate was defined as number of participants ≥18 years old with culture-confirmed TB disease (defined as positive culture for MTB) and those <18 years old with probable (clinical) TB disease (defined as objective evidence of clinical TB disease [cough, fever, night sweats, weight loss, or hemoptysis] based on history or physical exam plus radiograph, CT scan, other diagnostic tests PLUS response to antituberculosis therapy AND objective improvement of radiograph or other diagnostic tests; OR evidence of granuloma with organism positive for AFB], or caseating granulomata at autopsy or biopsy) between enrollment and 24 months after completion of study therapy per 100 participants with up to 33 months of follow-up and was calculated using survival analysis methods (Kaplan-Meier approach).
Time Frame: Baseline up to Month 27 (3RPT/INH) or Month 33 (9INH)
Population: MITT Population
Measure: Number; unit: TB cases per 100 participants w/followup
Groups:
- 9INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV infected participants) self-administered oral INH tablets (aged ≥12 years of age received 5 mg/kg and participants 2-11 years of age received 10-15 mg/kg) once daily for 9 months (240 to 270 total doses).
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 3651 | 3914
TB cases per 100 participants w/followup | 0.37 | 0.16
Statistical Analysis 1: Comparison: 9INH vs 3RPT/INH; Test type: Non-Inferiority or Equivalence — The noninferiority test statistic was based on the difference of the nonparametric Kaplan-Meier estimators. The asymptotic variance of the test statistic was obtained through Greenwood's formula and a two-sided 95% CI was constructed for the difference. If the upper bound of the CI was smaller than the noninferiority margin 0.75%, then the null hypothesis would be rejected and noninferiority could be claimed; Difference in Cumulative TB Rate = -0.21, 95% CI 1-sided [upper limit 0.04] — The difference in cumulative TB disease rate is the percentage in the 3RPT/INH arm minus the percentage in the 9INH arm

3. Secondary Outcome: Cumulative Rate of Culture-Confirmed or Probable (Clinical) TB Disease (Regardless of Age) At 33 Months After Enrollment
Description: Cumulative TB disease rate was defined as number of participants (regardless of age) with culture-confirmed TB disease (defined as positive culture for MTB]) or probable (clinical) TB disease (defined as objective evidence of clinical TB disease [cough, fever, night sweats, weight loss, or hemoptysis] based on history or physical exam plus radiograph, CT scan, other diagnostic tests PLUS response to antituberculosis therapy AND objective improvement of radiograph or other diagnostic tests; OR evidence of granuloma with organism positive for AFB, or caseating granulomata at autopsy or biopsy) between enrollment and the 990th Day of the Trial (33 months after enrollment, or end of the trial) per 100 participants w/33 months of follow-up and was calculated using survival analysis methods (Kaplan-Meier approach).
Time Frame: Baseline up to 33 Months
Measure: Number; unit: TB cases per 100 participants w/followup
Groups:
- 9INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR], HIV infected participants) self-administered oral INH tablets (aged ≥12 years of age received 5 mg/kg and participants 2-11 years of age received 10-15 mg/kg) once daily for 9 months (240 to 270 total doses).
- 3RPT/INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV-infected participants) received oral INH tablets (≥12 years of age received 15 mg/kg and participants 2-11 years of age received 25 mg/kg) and oral RPT tablets (between 300-900 mg based on weight) once per week for 3 months (11 to 12 total doses) administered by DOT, defined as a healthcare worker observing ingestion of each dose of RPT and INH.
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 3745 | 3986
TB cases per 100 participants w/followup | 0.49 | 0.24
Statistical Analysis 1: Comparison: 9INH vs 3RPT/INH; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in Cumulative TB Disease Rate = -0.25, 95% CI 1-sided [upper limit 0.03] — The difference in cumulative TB disease rate is the percentage in the 3RPT/INH arm minus the percentage in the 9INH arm

4. Secondary Outcome: Percentage of Participants With Drug Discontinuation Due to Adverse Drug Reactions Associated With 3RPT/INH or 9INH
Description: Discontinuation of study drug due to an adverse drug reaction associated with either 3RPT/INH or 9INH was defined as discontinuing treatment and/or study due to a treatment-related adverse event (AE) (considered either possibly, probably, or definitely related to the study drug by the investigator).
Time Frame: Baseline up to 60 days after the last dose of study drug (Month 5 [3RPT/INH] or Month 11 [9INH])
Population: Safety Population: all participants who enrolled in the study and took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 3759 | 4040
percentage of participants | 3.8 | 4.9
Statistical Analysis 1: Comparison: 9INH vs 3RPT/INH; Test type: Superiority or Other; p = 0.02, Chi-squared

5. Secondary Outcome: Percentage of Patients With Grade 3 or 4 Drug Toxicities Associated With 3RPT/INH or 9INH
Description: Drug toxicities (or AEs) were graded using Common Toxicity Criteria (CTC version 2.0, Publish Date April 30, 1999, Cancer Therapy Evaluation Program). Grade 3 and 4 drug toxicities associated with 3RPT/INH or 9INH were defined as treatment-related Grade 3 or 4 AEs (considered either possibly, probably, or definitely related to the study drug by the investigator).
Time Frame: Baseline up to 60 days after the last dose of study drug (Month 5 [3RPT/INH] or Month 11 [9INH])
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 3759 | 4040
percentage of participants
  Grade 3 | 2.2 | 2.7
  Grade 4 | 0.4 | 0.4
Statistical Analysis 1: Comparison: 9INH vs 3RPT/INH; Grade 3 Drug Toxicity; Test type: Superiority or Other; p = 0.24, Chi-squared
Statistical Analysis 2: Comparison: 9INH vs 3RPT/INH; Grade 4 Drug Toxicity; Test type: Superiority or Other; p = 0.59, Chi-squared

6. Secondary Outcome: Percentage of Participants With Death Due to Any Cause
Time Frame: Baseline up to Month 35
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 3759 | 4040
percentage of participants | 1.0 | 0.8
Statistical Analysis 1: Comparison: 9INH vs 3RPT/INH; Test type: Superiority or Other; p = 0.22, Chi-squared

7. Secondary Outcome: Percentage of Participants With Methadone Withdrawal Associated With 3RPT/INH and 9INH Among Participants Receiving Concomitant Methadone
Description: Among participants concomitantly receiving methadone, the development of methadone withdrawal (defined as having >3 new symptoms for >7 days: nausea and vomiting, abdominal cramps, body aches, restlessness, irritability, dilated pupils, tremors, involuntary twitching, lacrimation, rhinorrhea, sneezing, yawning, excessive perspiration, goose flesh, or diarrhea).
Time Frame: Baseline to Month 33
Measure: Count of Participants; unit: Participants
Groups:
- 9INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV infected participants) self-administered oral INH tablets (participants receiving concomitant methadone) once daily for 9 months daily self- administered isoniazid, 5mg/kg (300 mg max; 240 to 270 total doses).
- 3RPT/INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV-infected participants) (participants receiving concomitant methadone) received oral INH tablets (15 mg/kg; 900 mg max) and oral RPT tablets (between 300-900 mg based on weight) once per week for 3 months (11 to 12 total doses) administered by DOT, defined as a healthcare worker observing ingestion of each dose of RPT and INH.
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 77 | 75
Participants | 14 | 15

8. Secondary Outcome: Percentage of Participants With Drug Discontinuation for Any Reason Associated With 3RPT/INH or 9INH
Description: Drug discontinuations for any reason associated with 3RPT/INH or 9INH included all reasons for discontinuation from study treatment, regardless of relationship to treatment.
Time Frame: Baseline up to Month 3 (3RPT/INH) or Month 9 (9INH)
Population: MITT Population
Measure: Number; unit: percentage of participants
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 3745 | 3986
percentage of participants | 31.0 | 17.9
Statistical Analysis 1: Comparison: 9INH vs 3RPT/INH; Test type: Superiority or Other; p < 0.001, Chi-squared

9. Secondary Outcome: Percentage of Participants Who Completed the Treatment Regimen
Description: Completion in the 3RPT/INH arm was defined as: received 12 doses of RPT/INH within 16 weeks (12 weeks optimal). However, participants were considered to have completed therapy if at least 11 doses of RPT/INH had been received (~90%) during the 16-week time period. Completion in the 9INH arm was defined as: received 270 doses of INH within 52 weeks (39 weeks optimal). However, participants were considered to have completed therapy if at least 240 doses of INH were received (~90%) during the 52-week period.
Time Frame: Baseline up to Month 3 (3RPT/INH) or Month 9 (9INH)
Population: MITT Population
Measure: Number; unit: percentage of participants
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 3745 | 3986
percentage of participants | 69.0 | 82.1
Statistical Analysis 1: Comparison: 9INH vs 3RPT/INH; Test type: Superiority or Other; p < 0.0001, Chi-squared

10. Secondary Outcome: Cumulative Rate of Culture-Confirmed TB Disease in Participants ≥18 Years of Age AND Culture Confirmed or Probable (Clinical) TB Disease Among Participants <18 Years of Age Who Completed Study Phase Therapy Within 33 Months of Enrollment
Description: Cumulative TB disease rate was defined as number of participants ≥18 years old with culture-confirmed TB disease (defined as positive culture for MTB) and <18 years old with probable (clinical) TB disease (defined as objective evidence of clinical TB disease [cough, fever, night sweats, weight loss, or hemoptysis] based on history or physical exam plus radiograph, CT scan, other diagnostic tests PLUS response to antituberculosis therapy AND objective improvement of radiograph or other diagnostic tests; OR evidence of granuloma with organism positive for AFB], or caseating granulomata at autopsy or biopsy) between enrollment and 33 months after enrollment (for those who completed therapy within 33 months) per 100 participants w/33 months of follow-up and was calculated using survival analysis methods (Kaplan-Meier approach).
Time Frame: Baseline up to Month 33
Population: Per Protocol Population: all enrolled and eligible participants (MITT Population) who completed study drug within targeted time period (11-12 3RPT/INH doses within 10-16 weeks; 240-270 INH doses within 35-52 weeks) or developed TB disease or died while on study therapy (or follow-up) but completed ≥75% of expected number of doses prior to event.
Measure: Number; unit: TB cases per 100 participants w/followup
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 2585 | 3273
TB cases per 100 participants w/followup | 0.11 | 0.05
Statistical Analysis 1: Comparison: 9INH vs 3RPT/INH; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in Cumulative TB Disease Rate = -0.19, 95% CI 1-sided [upper limit 0.06] — The difference in cumulative TB disease rate is the percentage in the 3RPT/INH arm minus the percentage in the 9INH arm

11. Secondary Outcome: Percentage of Participants With Resistance to Study Medications in Isolates of MTB From Participants Who Developed Active TB Disease Within 33 Months of Enrollment
Description: Drug-susceptibility testing (DST) was performed on isolates of MTB obtained from participants who developed signs and symptoms of active TB disease (including sputum specimens or specimens from appropriate body site for extrapulmonary TB disease). DST was performed at site's local laboratory and sent to Sponsor for confirmatory susceptibility testing. DST included all drugs currently used to treat TB disease, including pyrazinamide (PZA) and fluoroquinolones. Susceptibility was tested for other drugs at the Sponsor laboratory at the following concentrations: INH, 0.02, 1.0, and 5.0 micrograms per milliliter (µg/mL) and rifampin (RIF), 1.0 µg/mL. Isolates resistant to RIF were assumed to be resistant to RPT.
Time Frame: Baseline up to Month 33
Population: N equals the number of participants who developed active TB disease during the study for which DST was performed.
Measure: Number; unit: percentage of participants
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 13 | 7
percentage of participants
  INH monoresistance | 15 | 0
  RIF and PZA resistant | 0 | 14

12. Secondary Outcome: Cumulative Rate of Culture-Confirmed or Probable TB Disease in HIV-Infected Participants Within 33 Months After Enrollment
Description: Cumulative TB disease rate was defined as number of HIV-infected participants ≥2 years old with culture-confirmed TB disease (defined as positive culture for MTB) or probable (clinical) TB disease (defined as objective evidence of clinical TB disease [cough, fever, night sweats, weight loss, or hemoptysis] based on history or physical exam plus radiograph, CT scan, other diagnostic tests PLUS response to antituberculosis therapy AND objective improvement of radiograph or other diagnostic tests; OR evidence of granuloma with organism positive for AFB], or caseating granulomata at autopsy or biopsy) between enrollment and the 990th day of the trial (33 months after enrollment, or end of the trial) per 100 participants w/33 months of follow-up and was calculated using survival analysis methods (Kaplan-Meier approach).
Time Frame: Baseline to Month 33
Measure: Number; unit: TB cases per 100 participants w/followup
Groups:
- 9INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV infected participants) self-administered oral INH tablets (HIV infected participants) once daily for 9 months daily self- administered isoniazid, 5mg/kg (300 mg max; 240 to 270 total doses).
- 3RPT/INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV-infected participants) (HIV infected participants) received oral INH tablets (15 mg/kg; 900 mg max) and oral RPT tablets (between 300-900 mg based on weight) once per week for 3 months (11 to 12 total doses) administered by DOT, defined as a healthcare worker observing ingestion of each dose of RPT and INH.
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 193 | 206
TB cases per 100 participants w/followup | 3.5 | 1.01

13. Secondary Outcome: Cumulative Rate of HIV-Infected Participants With Culture-Confirmed or Probable TB Disease at 24 Months After Completion of Study Therapy
Description: Cumulative TB disease rate was defined as number of HIV-infected participants with culture-confirmed TB (defined as positive culture for MTB) or probable (clinical) TB disease (defined as objective evidence of clinical TB disease [cough, fever, night sweats, weight loss, or hemoptysis] based on history or physical exam plus radiograph, CT scan, other diagnostic tests PLUS response to antituberculosis therapy AND objective improvement of radiograph or other diagnostic tests; OR evidence of granuloma with organism positive for AFB], or caseating granulomata at autopsy or biopsy) between enrollment and 24 months after completion of study therapy per 100 participants with up to 33 months of follow-up and was calculated using survival analysis methods (Kaplan-Meier approach).
Time Frame: Baseline up to Month 27 (3RPT/INH) or Month 33 (9INH)
Measure: Number; unit: TB cases per 100 participants w/followup
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 185 | 194
TB cases per 100 participants w/followup | 3.12 | 1.07

14. Secondary Outcome: Cumulative Rate of Participants <18 Years Old With Culture-Confirmed or Probable (Clinical) TB Disease Within 33 Months of Enrollment
Description: Cumulative TB disease rate was defined as number of participants <18 years old with culture-confirmed TB disease (defined as positive culture for MTB) or probable (clinical) TB disease (defined as objective evidence of clinical TB disease [cough, fever, night sweats, weight loss, or hemoptysis] based on history or physical exam plus radiograph, CT scan, other diagnostic tests PLUS response to antituberculosis therapy AND objective improvement of radiograph or other diagnostic tests; OR evidence of granuloma with organism positive for AFB], or caseating granulomata at autopsy or biopsy) between enrollment and the 990th day of the trial (33 months after enrollment, or end of the trial) per 100 participants w/33 months of follow-up and was calculated using survival analysis methods (Kaplan-Meier approach).
Time Frame: Baseline up to Month 33
Measure: Number; unit: TB cases per 100 participants w/followup
Groups:
- 9INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV infected participants) self-administered oral INH tablets (participants <18 years old) once daily for 9 months daily self- administered isoniazid, 5mg/kg (300 mg max; 240 to 270 total doses).
- 3RPT/INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV-infected participants) (participants <18 years old) received oral INH tablets (15 mg/kg; 900 mg max) and oral RPT tablets (between 300-900 mg based on weight) once per week for 3 months (11 to 12 total doses) administered by DOT, defined as a healthcare worker observing ingestion of each dose of RPT and INH.
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 434 | 471
TB cases per 100 participants w/followup | 0.74 | 0.00

15. Secondary Outcome: Cumulative Rate of Participants <12 Years Old With Culture-Confirmed or Probable (Clinical) TB Disease Within 33 Months of Enrollment
Description: Cumulative TB disease rate was defined as number of participants <12 years old with culture-confirmed TB disease (defined as positive culture for MTB) or probable (clinical) TB disease (defined as objective evidence of clinical TB disease [cough, fever, night sweats, weight loss, or hemoptysis] based on history or physical exam plus radiograph, CT scan, other diagnostic tests PLUS response to antituberculosis therapy AND objective improvement of radiograph or other diagnostic tests; OR evidence of granuloma with organism positive for AFB], or caseating granulomata at autopsy or biopsy) between enrollment and the 990th day of the trial (33 months after enrollment, or end of the trial) per 100 participants w/33 months of follow-up and was calculated using survival analysis methods (Kaplan-Meier approach).
Time Frame: Baseline up to Month 33
Measure: Number; unit: TB cases per 100 participants w/followup
Groups:
- 9INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV infected participants) self-administered oral INH tablets (participants <12 years old) once daily for 9 months daily self- administered isoniazid, 5mg/kg (300 mg max; 240 to 270 total doses).
- 3RPT/INH: Participants who were high-risk TST reactors (household and other close contacts of active TB cases, recent [within 2 years] tuberculin converters, participants with fibrotic lesions on CXR, HIV-infected participants) (participants <12 years old) received oral INH tablets (15 mg/kg; 900 mg max) and oral RPT tablets (between 300-900 mg based on weight) once per week for 3 months (11 to 12 total doses) administered by DOT, defined as a healthcare worker observing ingestion of each dose of RPT and INH.
Arm/Group | 9INH | 3RPT/INH
Number analyzed (Participants) | 178 | 234
TB cases per 100 participants w/followup | 1.35 | 0.00

ADVERSE EVENTS:
Time Frame: Baseline until Month 35
Arm/Group | 9INH | 3RPT/INH
Serious Adverse Events (participants affected / at risk) | 102/3759 | 60/4040
Other Adverse Events (participants affected / at risk) | 226/3759 | 248/4040
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 9INH (N=3759) | 3RPT/INH (N=4040)
Hernia repair (Surgical and medical procedures) | 3 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 2
Ankle operation (Surgical and medical procedures) | 1 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 1
Abdominal operation (Surgical and medical procedures) | 1 | 1
Abscess drainage (Surgical and medical procedures) | 0 | 1
Alcohol detoxification (Surgical and medical procedures) | 1 | 0
Angioplasty (Surgical and medical procedures) | 0 | 1
Arteriovenous graft (Surgical and medical procedures) | 0 | 1
Cardiac operation (Surgical and medical procedures) | 0 | 1
Endometriosis ablation (Surgical and medical procedures) | 1 | 0
Craniotomy (Surgical and medical procedures) | 0 | 1
Gallbladder operation (Surgical and medical procedures) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Internal fixation of fracture (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Open reduction of fracture (Surgical and medical procedures) | 1 | 0
Salivary gland resection (Surgical and medical procedures) | 1 | 0
Thyroidectomy (Surgical and medical procedures) | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0
Varicose vein operation (Surgical and medical procedures) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 3 | 2
Bronchitis (Infections and infestations) | 2 | 1
Appendicitis perforated (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Oesophageal irritation (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 3 | 1
Depression suicidal (Psychiatric disorders) | 2 | 0
Drug dependence (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0
Disorientation (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Substance abuse (Psychiatric disorders) | 0 | 1
Suicidal behavior (Psychiatric disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest pain (General disorders) | 7 | 2
Chest discomfort (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Drug withdrawal convulsions (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Thalamic infarction (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 1
Hypertensive crisis (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Gestational diabetes (Metabolism and nutrition disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 9INH (N=3759) | 3RPT/INH (N=4040)
Hypersensitivity (Immune system disorders) | 17 | 153
Medication error (Injury, poisoning and procedural complications) | 36 | 27
Hepatitis (Hepatobiliary disorders) | 110 | 24
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 69 | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No